CLINICAL TRIAL: NCT03695549
Title: Root Coverage After the Use of Coronally Advanced Flap With Advanced Platelet Rich Fibrin (A- PRF) Compared With Subepithelial Connective Tissue Graft in Management of Miller Class I and II Gingival Recession. A Randomized Clinical Trial
Brief Title: Evaluation of Root Coverage After the Use of Coronally Advanced Flap Either With Advanced Paltelet Rich Fibrin or Subepithilial Connective Tissue Graft in Treatment of Miller Class I and II Gingival Recession.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, heba samir, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: assistant lecturer
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Gingival Recession
Keywords: advanced platelet rich fibrin,A-PRF
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): CAF+ APRF
  Interventions: Procedure: CAF + (A-PRF)
- control (Active Comparator): CAF+SCTG
  Interventions: Procedure: CAF+SCTG

INTERVENTIONS:
Procedure: CAF + (A-PRF) — advanced platelet rich fibrin prepared by low speed centrfugation concept(LSCC) together with coronally advanced flap .
  Arms: intervention
Procedure: CAF+SCTG — cornally advanced flap plus subepithilial connective tissue graft harvested from the palate
  Arms: control

SUMMARY:
patients with Miller class I , II gingival recession will be divided into 2 groups (control, intervention).the control one will receive coronally advanced flap with subepithililal connective tissue graft harvested from the palate while the intervention one will have coronally advanced flap with advanced platelet rich fibrin(A-PRF).as it represent a new generation of platelet concentrate allow for better healing and root coverage results.

Null hypothesis: In patients with Miller class I and II gingival recession, there is no difference in amount of root coverage (mm) following the application of SCTG+A-PRF compared to CAF+SCTG.

DETAILED DESCRIPTION:
* Population (P): Patients with single Miller class I, II gingival recessions.
* Intervention (I): Coronally advanced flap (CAF) plus platelet rich fibrin (A-PRF).
* Comparator (C): Coronally advanced flap (CAF) plus subepithelial connective tissue graft (SCTG).
* Primary Outcome (O): Root coverage (mm).
* Time frame: 9 months.
* Study design: Randomized controlled clinical trial.
* Patients are to be selected from the outpatient clinic of the department of Oral Medicine and Periodontology-Cairo University

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients 18 years old and older both males and females.
* Good oral hygiene after phase I therapy.
* Miller's class I or II gingival recession.
* Not using antibiotics, steroids, chemotherapy or other medications that may modify results of the surgery and healing.
* Cooperative patients able and accept to come for follow up appointments

Exclusion Criteria:

* Pregnant or lactating females.
* Current Smokers.
* Patients with any systemic disease that may affect the periodontal healing.
* Teeth with endodontic treatment, buccal restoration or caries.
* Patients with poor oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
root coverage | 9 months
  measured in millimeter

SECONDARY OUTCOMES:
Gingival esthetics | 9 months
  Root coverage esthetic score
Recession width | 9 months
  measured in millimeter
Clinical attachment level | 9 months
  measured in millimeter
Width of keratinized gingiva | 9 months
  measured in millimeter
Probing depth | 9 months
  measured in millimeter
Gingival thickness | 9 months
  measured in millimeter
Post-operative pain | measured daily for the first 2 weeks post- operatively.
  Visual analog scale (VAS) Questionnaire
Patient Satisfaction | 9 months
  Post-Surgical Patient Satisfaction Questionnaire
Early wound healing | 1,2,4 weeks post- surgical
  Early wound healing index

CONTACTS AND LOCATIONS:
Overall Officials: Heba Samir Mhmoud, assistant lecturer, Principal Investigator — Cairo University; Manal M Hosny, professor, Study Director — Cairo University; Engi A Mahmoud, assistant professor, Study Chair — Cairo University